CLINICAL TRIAL: NCT02497014
Title: The European Bifurcation Club Left Main Study: A Randomised Comparison of Single Versus Dual Stent Implantation for Distal Left Main True Coronary Bifurcation Lesions
Brief Title: The European Bifurcation Club Left Main Study
Acronym: EBC MAIN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: European Cardiovascular Research Center (Network)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MED-03
Record Dates: First submitted 2015-07-01; First posted 2015-07-14 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Percutaneous Transluminal Coronary Angioplasty; Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 Stent (Experimental): Patients who are going to receive 1 stent in the main vessel and the side vessel will be treated with kissing ballon inflation
  Interventions: Device: 1 Stent
- 2 Stents (Experimental): Patients who are going to receive 2 stents in both vessels
  Interventions: Device: 2 Stents

INTERVENTIONS:
Device: 1 Stent — Stenting of main vessel should be undertaken with a wire jailed in the side vessel to preserve side vessel flow and access. Stent diameter should be chosen according to diameter of the main vessel immediately distal to the bifurcation. Distal left main should be dilated with a short non-compliant balloon. Side vessel should be rewired and a kissing balloon inflation should be undertaken. Balloon sizes should be according to the diameter of the main and side vessel with individual high pressure inflation followed by a final lower pressure kiss dilatation. Proximal stented portion in the left main coronary artery should be dilated to full expansion using either low pressure dilatation of the kissing balloon pair or a separate individual balloon. It is preferred that non-compliant balloons should be used to limit overstretching of vessels. In case of specific situations described in the protocol the operator may choose to implant a side vessel stent, using same process as described above.
  Arms: 1 Stent
Device: 2 Stents — Coronary guide wires should be passed to LAD and Cx/intermediate arteries respectively. One should be designated the main vessel and one should be designated the side vessel. The planned dual stent technique is at the discretion of the operator but should be one of culotte, minicrush, T or TAP. If a crush procedure is chosen, it should ideally be of the DK variety. Stent diameter should be chosen according to the diameter of the vessel immediately distal to the bifurcation. Wire jail, POT, non-compliant balloons, high pressure individual "ostial" dilatations and final dilatation of the stented proximal left main should be used in accordance with the advice of the EBC. Further treatment to proximal or distal aspects of the main vessel or side vessel can be continued at the discretion of the operator. At any stage, proximal or distal dissections may be treated as required with further stent implantations. At any stage, post-dilatations may be undertaken to optimise stent expansion.
  Arms: 2 Stents

SUMMARY:
The objective of the study is to investigate clinical outcomes following single versus dual stenting strategies for the treatment of true bifurcation distal left main coronary artery lesions.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet ALL of the inclusion criteria:

* Bifurcation distal left main stem stenosis >50% and

  * Ischaemic symptoms, or
  * Positive non-invasive imaging for ischaemia, or
  * Positive FFR, or
  * LMS IVUS MLA <6mm2
* Left main diameter ≤5.75mm
* True bifurcation lesion type 1,1,1 or 0,1,1
* LAD and Cx diameter both >2.75mm
* Unprotected left main
* Patient ≥18 years old

Exclusion Criteria:

* STEMI <72 hours preceding
* Cardiogenic shock
* Chronic total occlusion of either vessel
* >2 other coronary lesions planned for treatment
* SYNTAX score for planned lesions to be treated >32
* LMS trifurcation if all vessels are ≥2.75mm diameter
* Either bifurcation vessel not suitable for stenting
* Platelet count ≤50 x 10^9/mm3
* Left ventricular ejection fraction ≤20%
* Patient life expectancy less than 12 months
* Participation in another investigational drug or device study
* Patient unable to give informed consent
* Women of child-bearing potential or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2016-02; Primary Completion 2018-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Composite of Death, Myocardial infarction and Target Lesion Revascularisation | 1 year

SECONDARY OUTCOMES:
Death | 1 year
Myocardial Infarction | 1 year
Target Lesion Revascularization | 1 year
Angina status | 1 year
Stent thrombosis | 1 year
Death | 3 years
Myocardial Infarction | 3 years
Target Lesion Revascularization | 3 years

OTHER OUTCOMES:
Procedure success by assessing a composite of the number of guidewires, balloons and stents opened or used and procedural time. | up to 18 months
Technical success by assessing a composite of the number of guidewires, balloons and stents opened or used and procedural time. | up to 18 months
Number of procedural and in-hospital Major adverse Cardiac Events (MACE) | up to 18 months
Procedure duration | intraoperative
Fluoroscopy by assessing a composite of the number of guidewires, balloons and stents opened or used and procedural time | up to 18 months
X-ray dose | up to 18 months
Economic evaluation by assessing all procedural costs for each stenting strategy | up to 18 months

CONTACTS AND LOCATIONS:
Overall Officials: David Hildick-Smith, Dr, Principal Investigator — Brighton and Sussex University Hospitals NHS Trust
Locations (24):
- Denmark (2):
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet Copenhagen University Hospital, Copenhagen
- France (6):
  - Clinique de Fontaine, Fontaine-lès-Dijon
  - HCL CHU Luis Pradel, Lyon
  - Hopital Jacques Cartier, Massy
  - Clinique Saint Hilaire, Rouen
  - Clinique Pasteur, Toulouse
  - CHU Rangueil, Toulouse
- Germany (2):
  - Herzzentrum Bad Krozingen, Bad Krozingen
  - Elisabeth Krankenhaus Essen, Essen
- Italy (3):
  - University of Catania - Ferrarotto Hospital, Catania
  - Ospedale San Raffaele, Milan
  - Universita Cattolica del Sacre Cuore, Roma
- Pauls Stradins Clinical University Hospital, Riga, Latvia
- Clinical Center of Serbia, Belgrade, Serbia
- Spain (4):
  - Hospital del Mar, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Sant Pau i Sant Creu, Barcelona
  - Hospital de la Reina Sofia, Córdoba
- United Kingdom (5):
  - Belfast City Hospital, Belfast
  - Royal Sussex County Hospital, Brighton
  - St Thomas Hospital, London
  - Freeman Hospital, Newcastle upon Tyne
  - John Radcliffe Hospital, Oxford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maznyczka A, Arunothayaraj S, Banning AP, Schmitz T, Wlodarczak A, Silvestri M, Egred M, Koning R, Spence MS, Morice MC, Lefevre T, Ferenc M, Cockburn J, Erglis A, Brunel P, Burzotta F, Kretov E, Hovasse T, Pan M, Clesham G, Chieffo A, Mylotte D, Lindsay M, Christiansen EH, Bouisset F, Vaquerizo B, Lassen JF, Darremont O, Louvard Y, Stankovic G, Hildick-Smith D; EBC MAIN (European Bifurcation Club Left Main Coronary Stent) Trial Investigators. Patterns of Restenosis After Left Main Bifurcation Single- or Dual-Stenting: An EBC MAIN Trial Subanalysis. Circ Cardiovasc Interv. 2025 Nov;18(11):e015546. doi: 10.1161/CIRCINTERVENTIONS.125.015546. Epub 2025 Sep 17. PMID 40959874
- [Derived] Arunothayaraj S, Egred M, Banning AP, Brunel P, Ferenc M, Hovasse T, Wlodarczak A, Pan M, Schmitz T, Silvestri M, Erglis A, Kretov E, Lassen JF, Chieffo A, Lefevre T, Burzotta F, Cockburn J, Darremont O, Stankovic G, Morice MC, Louvard Y, Hildick-Smith D. Stepwise Provisional Versus Systematic Dual-Stent Strategies for Treatment of True Left Main Coronary Bifurcation Lesions. Circulation. 2025 Mar 4;151(9):612-622. doi: 10.1161/CIRCULATIONAHA.124.071153. Epub 2025 Feb 5. PMID 39907022
- [Derived] Arunothayaraj S, Lassen JF, Clesham GJ, Spence MS, Koning R, Banning AP, Lindsay M, Christiansen EH, Egred M, Cockburn J, Mylotte D, Brunel P, Ferenc M, Hovasse T, Wlodarczak A, Pan M, Silvestri M, Erglis A, Kretov E, Chieffo A, Lefevre T, Burzotta F, Darremont O, Stankovic G, Morice MC, Louvard Y, Hildick-Smith D. Impact of technique on bifurcation stent outcomes in the European Bifurcation Club Left Main Coronary Trial. Catheter Cardiovasc Interv. 2023 Feb;101(3):553-562. doi: 10.1002/ccd.30575. Epub 2023 Jan 29. PMID 36709485
- [Derived] Hildick-Smith D, Egred M, Banning A, Brunel P, Ferenc M, Hovasse T, Wlodarczak A, Pan M, Schmitz T, Silvestri M, Erglis A, Kretov E, Lassen JF, Chieffo A, Lefevre T, Burzotta F, Cockburn J, Darremont O, Stankovic G, Morice MC, Louvard Y. The European bifurcation club Left Main Coronary Stent study: a randomized comparison of stepwise provisional vs. systematic dual stenting strategies (EBC MAIN). Eur Heart J. 2021 Oct 1;42(37):3829-3839. doi: 10.1093/eurheartj/ehab283. PMID 34002215